CLINICAL TRIAL: NCT03314025
Title: Prophylactic Tamsulosin in Prevention of Post-operative Urinary Retention in Men After Transanal Endoscopic Microsurgery: A Multicenter Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Prophylactic Tamsulosin in Prevention of Post-operative Urinary Retention in Men After Transanal Endoscopic Microsurgery
Acronym: TEMPOUR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015-2392
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention | interventions — Tamsulosin; Sugars

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everyone is blinded except the pharmacy department where the randomization list is kept. This department is the one able to unblind a patient, if needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin (Experimental): The patients in the Experimental group will receive Tamsulosin Hydrochloride 0.4 MG (milligrams) once a day for 5 days before the surgery, one capsule on the day of the surgery and one on the day after. The intervention will consist of a total of 7 capsules
  Interventions: Drug: Tamsulosin Hydrochloride 0.4 MG; Device: Foley catheter
- Placebo (Placebo Comparator): The patients in the Placebo group will receive a placebo oral capsule (sugar) once a day for 5 days before the surgery, one capsule on the day of the surgery and one on the day after. The intervention will consist of a total of 7 capsules
  Interventions: Drug: Placebo oral capsule; Device: Foley catheter

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride 0.4 MG — Peri-operative therapy of Tamsulosin Hydrochloride 0.4 milligrams daily for a total of 7 days.
  Other Names: Tamsulosin
  Arms: Tamsulosin
Drug: Placebo oral capsule — Peri-operative therapy of a Placebo oral capsule daily for a total of 7 days.
  Other Names: Sugar pill; Control
  Arms: Placebo
Device: Foley catheter — Every patient with a post-operative urinary retention will have a foley catheter, as standard of care.

SUMMARY:
Post-operative urinary retention (POUR) is a frequent complication reported as ranging from 10 to 55% in the literature. In a recent retrospective study from Laliberte et al in Quebec City, we observed that 19% of the patients operated using transanal endoscopic microsurgery (TEM) had a post-operative urinary retention (POUR). Factors related to the patient, the tumor and the surgery were not observed to be associated risk factors. Tamsulosin has been shown as an effective preventive agent of POUR for certain ano-rectal and inguinal surgeries. The efficacy of this prophylactic therapy in transanal endoscopic microsurgery has not been studied yet and is unclear considering the particularities of this procedure. TEM uses a rigid proctoscope of four centimeters of diameter and creates a continuous pneumorectum (insufflation of the rectum during all the procedure). We think that these two elements, which cause local inflammation, may be part of the reason explaining the high incidence of post-operative urinary retention after TEM procedures. The objective of our multicenter clinical trial is to evaluate the effect of perioperative tamsulosin for the reduction of POUR in men, as well as the impact on the interventions and hospital admissions related to this complication.

DETAILED DESCRIPTION:
We are conducting a feasibility study (Vanguard phase) with three Canadian centers :

1. CHU de Quebec - Laval University, Quebec City, Quebec, Canada
2. St-Paul's Hospital, Vancouver, British-Columbia, Canada
3. Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

Other Canadian centers will be offered to join our study if the Vanguard phase demonstrates the feasibility of this clinical trial.

Large scale study

We anticipate the detection of a 15% absolute risk reduction of POUR in the Experimental group in comparison with the Placebo group. To detect a 15% reduction of POUR in the Experimental group (10% anticipated) in comparison with the Placebo group (25% anticipated) and to assure a study power of 80% with a unilateral Chi2 and a significance level of 5%, we need 158 patients in total; 79 in each group.

Feasibility study (Vanguard phase)

We expect at least a 60% recruitment rate throughout the two first participating Canadian centers, which translates into a mean of 8 patients recruited each month overall. Regarding the medication adherence, two studies that evaluated the use patterns and adherence to medications for lower urinary tract symptoms suggestive of benign prostatic hyperplasia found an adherence of 67% to 89%, with a mean of 78%. Based on these two studies, we expect that the patients will at least take 80% of the medication at study. To detect an 80% medication adherence with a 95% confidence interval, we need 62 enrolled patients.

The research pharmacy at the CHU de Quebec - Laval University will be responsible for preparing the study drug. The active medication or the placebo (sugar) will be encapsulated using identical capsules. The research pharmacy at the coordinating center will provide the study drug and the placebo to the other participating centers. There will be a quality control of the capsules; a temperature monitor will be in the boxes sent to the other centers and a control on the expiration date will be made. The capsules that are not used will be destroyed at each center. The randomization will be kept at the CHU de Quebec - Laval University research center. Patients will be stratified by center.

The patients are asked to report any potential adverse effect and our data safety monitoring board will meet annually to assess these or sooner if any adverse effect is serious.

We justify the duration of the intervention by the time needed to reach a steady state, which is estimated to be 4 to 5 days. The 7-day therapy is also based on the study from Patel et al, which showed a significant reduction of acute urinary retention with a 7-day intake of tamsulosin. It is the common and recommended dose used in other patient population.

Data collection

Patients will be identified by a study number in the study database. A master list of participants linking their study number with their medical record number will be kept in the computer of the PI at every research center participating in the study, and will be password protected. Data will be collected prospectively at the bedside during the study period.

Statistical analysis

First, a descriptive analysis of the population at study will be performed for socio- demographic, anthropometric and clinical characteristics. The means, standard deviations, medians and interquartile ranges will be presented as continuous numerical variables, while the frequencies and percentages will be determined for categorical variables. In the large-scale study, a Chi-square test or Fisher Exact test, if appropriate, will be used for the analysis of the primary endpoint, which is the comparison of the rate of POUR in the Experimental group with the rate of POUR in the Placebo group. This same test will also be helpful in the analysis of the secondary endpoints. If the patient doesn't take all of his medication or his surgery is cancelled he will still be included, since this will be an intention-to-treat analysis. Sub-group analyses will be performed to evaluate the impact of the tumour's characteristics, the duration of the surgery, the volume of intravenous fluids received during the intervention, the type of anaesthesia and the International Prostate Symptom Score (IPSS).

Potential conflicts of interest

This is an investigator-led study that is independent and not sponsored by the industry. The study is funded through local funds (CHU de Quebec - Laval University, Department of Surgery) as well as from in-kind funding of the institution.

ELIGIBILITY:
Inclusion Criteria:

* Male patients of 18 years and older that are scheduled for a TEM resection during the study period.

Exclusion Criteria:

* Patient already taking an alpha1-adrenergic blocking agent Flomax® (Tamsulosin), Cardura® (Doxazosin), Hytrin® (Terazosine) Rapaflo® (Silodosin), Xatral® (Alfuzosin), Minipress® (Prazosin)
* Patient having an indwelling bladder catheter
* Allergy or hypersensibility to any alpha1-adrenergic blocking agent
* Patient taking one of the following:

Anti-retroviral therapy, Antifungal drug, Clarithromycin, Erythromycin, Paroxetine, Terbinafine, Cimetidine, Warfarin, Sildenafil, Tadalafil, Vardenafil (these drugs have possible interactions with the study drug)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Urinary Retention (POUR) (yes or no) | 6 hours
  The absence of natural voiding after a surgery needing an intervention as a Foley catheter or a catheterization. If the patient needs this intervention, he will be stated to have had a POUR.

SECONDARY OUTCOMES:
Side effects of Tamsulosin Hydrochloride | 7 days
  Every potential side effect will be reported
Hospital admission | 24 hours
  Every admission related to the primary outcome
Indwelling catheter | 1 month
  Duration of the indwelling catheter (24-48 hours vs more than 48 hours)
Recurrence | 24 hours after the removal of the catheter
  Recurrence of urinary retention after catheter removal
The International Prostate Symptom Score (IPSS) Score | 7 days
  The standardized questionnaire will be submitted to the patients before and after the prophylactic therapy. The score is out of 35.
  Score Correlation
  0-7 Mildly symptomatic
  8-19 Moderately symptomatic
  20-35 Severely symptomatic
Late POUR | Between 6 hours and 24 hours post-op
  Late post-operative urinary retention

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Drolet, MD FRCSC, Principal Investigator — CHU de Quebec-Universite Laval
Locations (3):
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - CHU de Quebec - Universite Laval, Québec, Quebec

REFERENCES:
- [Background] Akkoc A, Aydin C, Topaktas R, Kartalmis M, Altin S, Isen K, Metin A. Prophylactic effects of alpha-blockers, Tamsulosin and Alfuzosin, on postoperative urinary retention in male patients undergoing urologic surgery under spinal anaesthesia. Int Braz J Urol. 2016 May-Jun;42(3):578-84. doi: 10.1590/S1677-5538.IBJU.2015.0256. PMID 27286124
- [Background] Bailey HR, Ferguson JA. Prevention of urinary retention by fluid restriction following anorectal operations. Dis Colon Rectum. 1976 Apr;19(3):250-2. doi: 10.1007/BF02590913. PMID 1269351
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Background] Barkin J, Diles D, Franks B, Berner T. Alpha blocker monotherapy versus combination therapy with antimuscarinics in men with persistent LUTS refractory to alpha-adrenergic treatment: patterns of persistence. Can J Urol. 2015 Aug;22(4):7914-23. PMID 26267031
- [Background] Bozlu M, Ulusoy E, Doruk E, Cayan S, Canpolat B, Schellhammer PF, Akbay E. Voiding impairment after prostate biopsy: does tamsulosin treatment before biopsy decrease this morbidity? Urology. 2003 Dec;62(6):1050-3. doi: 10.1016/j.urology.2003.07.006. PMID 14665353
- [Background] Buckley BS, Lapitan MC. Drugs for treatment of urinary retention after surgery in adults. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD008023. doi: 10.1002/14651858.CD008023.pub2. PMID 20927768
- [Background] Cataldo PA, Senagore AJ. Does alpha sympathetic blockade prevent urinary retention following anorectal surgery? Dis Colon Rectum. 1991 Dec;34(12):1113-6. doi: 10.1007/BF02050073. PMID 1959461
- [Background] Chung SJ, Jung SI, Ryu JW, Hwang EC, Kwon DD, Park K, Kim JW. The preventive effect of tamsulosin on voiding dysfunction after prostate biopsy: a prospective, open-label, observational study. Int Urol Nephrol. 2015 May;47(5):711-5. doi: 10.1007/s11255-015-0955-7. Epub 2015 Mar 27. PMID 25812823
- [Background] Dreijer B, Moller MH, Bartholdy J. Post-operative urinary retention in a general surgical population. Eur J Anaesthesiol. 2011 Mar;28(3):190-4. doi: 10.1097/EJA.0b013e328341ac3b. PMID 21206278
- [Background] Elshaikh MA, Ulchaker JC, Reddy CA, Angermeier KW, Klein EA, Chehade N, Altman A, Ciezki JP. Prophylactic tamsulosin (Flomax) in patients undergoing prostate 125I brachytherapy for prostate carcinoma: final report of a double-blind placebo-controlled randomized study. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):164-9. doi: 10.1016/j.ijrobp.2004.09.036. PMID 15850917
- [Background] Fisher E, Subramonian K, Omar MI. The role of alpha blockers prior to removal of urethral catheter for acute urinary retention in men. Cochrane Database Syst Rev. 2014 Jun 10;2014(6):CD006744. doi: 10.1002/14651858.CD006744.pub3. PMID 24913721
- [Background] Goldman G, Leviav A, Mazor A, Kashtan H, Aladgem D, Greenstein A, Wiznitzer T. Alpha-adrenergic blocker for posthernioplasty urinary retention. Prevention and treatment. Arch Surg. 1988 Jan;123(1):35-6. doi: 10.1001/archsurg.1988.01400250037005. PMID 3337653
- [Background] Gonullu NN, Dulger M, Utkan NZ, Canturk NZ, Alponat A. Prevention of postherniorrhaphy urinary retention with prazosin. Am Surg. 1999 Jan;65(1):55-8. PMID 9915533
- [Background] Jang JH, Kang SB, Lee SM, Park JS, Kim DW, Ahn S. Randomized controlled trial of tamsulosin for prevention of acute voiding difficulty after rectal cancer surgery. World J Surg. 2012 Nov;36(11):2730-7. doi: 10.1007/s00268-012-1712-z. PMID 22806208
- [Background] Jeong IG, You D, Yoon JH, Hong S, Lim JH, Hong JH, Choo MS, Ahn H, Kim CS. Impact of tamsulosin on urinary retention following early catheter removal after robot-assisted laparoscopic radical prostatectomy: a prospective randomized controlled trial. Int J Urol. 2014 Feb;21(2):164-8. doi: 10.1111/iju.12225. Epub 2013 Jul 30. PMID 23906190
- [Background] Jordan CG. Post-Operative Urinary Retention. Ann Surg. 1933 Jul;98(1):125-37. doi: 10.1097/00000658-193307000-00012. No abstract available. PMID 17867002
- [Background] Kapoor A. Benign prostatic hyperplasia (BPH) management in the primary care setting. Can J Urol. 2012 Oct;19 Suppl 1:10-7. PMID 23089343
- [Background] Keita H, Diouf E, Tubach F, Brouwer T, Dahmani S, Mantz J, Desmonts JM. Predictive factors of early postoperative urinary retention in the postanesthesia care unit. Anesth Analg. 2005 Aug;101(2):592-596. doi: 10.1213/01.ANE.0000159165.90094.40. PMID 16037182
- [Background] Lamonerie L, Marret E, Deleuze A, Lembert N, Dupont M, Bonnet F. Prevalence of postoperative bladder distension and urinary retention detected by ultrasound measurement. Br J Anaesth. 2004 Apr;92(4):544-6. doi: 10.1093/bja/aeh099. Epub 2004 Feb 20. PMID 14977795
- [Background] Laliberte AS, Lebrun A, Drolet S, Bouchard P, Bouchard A. Transanal endoscopic microsurgery as an outpatient procedure is feasible and safe. Surg Endosc. 2015 Dec;29(12):3454-9. doi: 10.1007/s00464-015-4158-1. Epub 2015 Mar 24. PMID 25801107
- [Background] Leventhal A, Pfau A. Pharmacologic management of postoperative overdistention of the bladder. Surg Gynecol Obstet. 1978 Mar;146(3):347-8. PMID 625669
- [Background] Livne PM, Kaplan B, Ovadia Y, Servadio C. Prevention of post-hysterectomy urinary retention by alpha-adrenergic blocker. Acta Obstet Gynecol Scand. 1983;62(4):337-40. doi: 10.3109/00016348309156234. PMID 6138916
- [Background] Lose G, Lindholm P. Prophylactic phenoxybenzamine in the prevention of postoperative retention of urine after vaginal repair: a prospective randomized double-blind trial. Int J Gynaecol Obstet. 1985 Sep;23(4):315-20. doi: 10.1016/0020-7292(85)90026-8. PMID 2866119
- [Background] Lowe FC. Summary of clinical experiences with tamsulosin for the treatment of benign prostatic hyperplasia. Rev Urol. 2005;7 Suppl 4(Suppl 4):S13-21. PMID 16986050
- [Background] Lucas MG, Stephenson TP, Nargund V. Tamsulosin in the management of patients in acute urinary retention from benign prostatic hyperplasia. BJU Int. 2005 Feb;95(3):354-7. doi: 10.1111/j.1464-410X.2005.05299.x. PMID 15679793
- [Background] Agrawal MS, Yadav A, Yadav H, Singh AK, Lavania P, Jaiman R. A prospective randomized study comparing alfuzosin and tamsulosin in the management of patients suffering from acute urinary retention caused by benign prostatic hyperplasia. Indian J Urol. 2009 Oct-Dec;25(4):474-8. doi: 10.4103/0970-1591.57917. PMID 19955671
- [Background] Madani AH, Aval HB, Mokhtari G, Nasseh H, Esmaeili S, Shakiba M, Shakiba RS, Seyed Damavand SM. Effectiveness of tamsulosin in prevention of post-operative urinary retention: a randomized double-blind placebo-controlled study. Int Braz J Urol. 2014 Jan-Feb;40(1):30-6. doi: 10.1590/S1677-5538.IBJU.2014.01.05. PMID 24642148
- [Background] Mason SE, Scott AJ, Mayer E, Purkayastha S. Patient-related risk factors for urinary retention following ambulatory general surgery: a systematic review and meta-analysis. Am J Surg. 2016 Jun;211(6):1126-34. doi: 10.1016/j.amjsurg.2015.04.021. Epub 2015 Jul 17. PMID 26257154
- [Background] Mohammadi-Fallah M, Hamedanchi S, Tayyebi-Azar A. Preventive effect of tamsulosin on postoperative urinary retention. Korean J Urol. 2012 Jun;53(6):419-23. doi: 10.4111/kju.2012.53.6.419. Epub 2012 Jun 19. PMID 22741052
- [Background] Basheer A, Alsaidi M, Schultz L, Chedid M, Abdulhak M, Seyfried D. Preventive effect of tamsulosin on postoperative urinary retention in neurosurgical patients. Surg Neurol Int. 2017 May 10;8:75. doi: 10.4103/sni.sni_5_17. eCollection 2017. PMID 28584678
- [Background] Nasu K, Moriyama N, Fukasawa R, Tsujimoto G, Tanaka T, Yano J, Kawabe K. Quantification and distribution of alpha1-adrenoceptor subtype mRNAs in human proximal urethra. Br J Pharmacol. 1998 Apr;123(7):1289-93. doi: 10.1038/sj.bjp.0701731. PMID 9579721
- [Background] Patel R, Fiske J, Lepor H. Tamsulosin reduces the incidence of acute urinary retention following early removal of the urinary catheter after radical retropubic prostatectomy. Urology. 2003 Aug;62(2):287-91. doi: 10.1016/s0090-4295(03)00333-9. PMID 12893337
- [Background] Petersen MS, Collins DN, Selakovich WG, Finkbeiner AE. Postoperative urinary retention associated with total hip and total knee arthroplasties. Clin Orthop Relat Res. 1991 Aug;(269):102-8. PMID 1864026
- [Background] Petros JG, Bradley TM. Factors influencing postoperative urinary retention in patients undergoing surgery for benign anorectal disease. Am J Surg. 1990 Apr;159(4):374-6. doi: 10.1016/s0002-9610(05)81274-7. PMID 2316800
- [Background] Reitz A, Haferkamp A, Kyburz T, Knapp PA, Wefer B, Schurch B. The effect of tamsulosin on the resting tone and the contractile behaviour of the female urethra: a functional urodynamic study in healthy women. Eur Urol. 2004 Aug;46(2):235-40; discussion 240. doi: 10.1016/j.eururo.2004.04.009. PMID 15245819
- [Background] Shaw MK, Pahari H. The role of peri-operative use of alpha-blocker in preventing lower urinary tract symptoms in high risk patients of urinary retention undergoing inguinal hernia repair in males above 50 years. J Indian Med Assoc. 2014 Jan;112(1):13-4, 16. PMID 25935942
- [Background] Tammela T, Kontturi M, Puranen J. Prevention of postoperative urinary retention after total hip arthroplasty in male patients. Ann Chir Gynaecol. 1987;76(3):170-2. PMID 3314645
- [Background] Toyonaga T, Matsushima M, Sogawa N, Jiang SF, Matsumura N, Shimojima Y, Tanaka Y, Suzuki K, Masuda J, Tanaka M. Postoperative urinary retention after surgery for benign anorectal disease: potential risk factors and strategy for prevention. Int J Colorectal Dis. 2006 Oct;21(7):676-82. doi: 10.1007/s00384-005-0077-2. Epub 2006 Mar 22. PMID 16552523
- [Background] Verhamme KM, Dieleman JP, Bleumink GS, Bosch JL, Stricker BH, Sturkenboom MC. Treatment strategies, patterns of drug use and treatment discontinuation in men with LUTS suggestive of benign prostatic hyperplasia: the Triumph project. Eur Urol. 2003 Nov;44(5):539-45. doi: 10.1016/s0302-2838(03)00376-2. PMID 14572751
- [Background] Wu AK, Auerbach AD, Aaronson DS. National incidence and outcomes of postoperative urinary retention in the Surgical Care Improvement Project. Am J Surg. 2012 Aug;204(2):167-71. doi: 10.1016/j.amjsurg.2011.11.012. Epub 2012 May 3. PMID 22560203
- [Derived] Couture T, Morin C, Charbonneau J, Papillon-Dion E, Bouchard A, Rouleau-Fournier F, Bouchard P, Letarte F, Turgeon AF, Drolet S. TEMPOUR: A Randomized Controlled Trial Assessing Perioperative Use of an Alpha-1 Blocker to Reduce Postoperative Urinary Retention After Transanal Endoscopic Microsurgery Procedures. Dis Colon Rectum. 2025 Apr 1;68(4):475-482. doi: 10.1097/DCR.0000000000003623. Epub 2025 Jan 2. PMID 39745289